CLINICAL TRIAL: NCT02830958
Title: Postoperative Kinesio Taping Effect on Pain and Edema in Patients Who Underwent Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Kinesiotaping PTH
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Replacement, Total Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesiotaping Group (Experimental): applied next to the lymphatic system from the validated methods Kinesiotaping®.
  Interventions: Device: Kinesiotaping
- Ordinary tape Group (Placebo Comparator): Installation of an ordinary tape (not having the characteristics of Curetape®).
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Kinesiotaping — The Kinesio Taping® Method is a definitive rehabilitative taping technique that is designed to facilitate the body's natural healing process while providing support and stability to muscles and joints without restricting the body's range of motion as well as providing extended soft tissue manipulation to prolong the benefits of manual therapy administered within the clinical setting. Latex-free and wearable for days at a time, Kinesio® Tex Tape is safe for populations ranging from pediatric to geriatric, and successfully treats a variety of orthopedic, neuromuscular, neurological and other medical conditions.
  Arms: Kinesiotaping Group
Other: No intervention — No intervention. Uses of an ordinary tape
  Arms: Ordinary tape Group

SUMMARY:
The hip is a commonly performed operation corresponding to a prosthetic joint replacement surgery whose effectiveness depends on the quality of architectural and mechanical reconstruction of the artificial hip, integrity and balance of the periarticular musculature. To achieve this dual purpose, two elements are essential: access to the hip that best meets the musculature and is able to restore the balance, and adequate prosthesis. Despite the move towards a surgery less invasive hip replacement is a procedure that causes tissue damage. This results in nociceptive and neuropathic pain, which can become chronic in about 30% of cases.

Several studies have shown that there are risk factors for chronic post-surgical pain. They are both related to patients but also to surgery. It is thus advantageous to reduce the postoperative pain, localized mainly in the trochanteric region, to decrease the risk of developing chronic post surgical pain. Now medical comunity know that the post-operative bruising and tissue damage are partly responsible for these pains.

The Kinesiotaping uses an adhesive elastic cotton tape color invented by Dr. Kase in the 1970s It is water resistant and retains its properties up to 5 days. It has the characteristic to cause elevation of the epidermis and thereby reduce the pressure on the mechanoreceptors below the dermis. This would have the effect of reducing nociceptive stimuli.

Its designers also claim it would have a beneficial effect on the lymphatic and venous circulation. According Kase Kinesiotaping causes an uprising of the epidermis decreasing the pressure in the dermis and promoting lymphatic drainage through its mechanical action during movement.

The lymphatic system is responsible for the capture of waste from venous blood (catabolites, plasma proteins) and thus can promote the absorption of edema.

In his study, Donec highlights a significant decrease in pain and a higher absorption of postoperative edema in the Kinésiotape® group than in the control group in surgical patients with total knee arthroplasty .

The Curetape® band is used in the orthopedic surgery department since 2010 in current care.

Consequently, it seems interesting to evaluate the effect of Curetape® in surgical patients with a total hip replacement.

DETAILED DESCRIPTION:
Main objectives / Secondary:

To evaluate the effect of the application of Kinésiotape® in patients undergoing a total hip replacement on pain and changes in the immediate postoperative edema.

Methodology :

* STUDY This will be a prospective randomized study in routine care, against placebo performed in the hospital group Paris Saint Joseph, 75014.
* Randomization:

Given the weakness of the literature on this subject Investigators opted for a trial randomization into 2 groups that will be made by the patient. The patient list will be balanced by randomly alternating blocks. the orthopedic ward staff and physiotherapists will not be informed of the first schedule to avoid a bias in the care of patients. An array of randomization will be created by an independent person in the study. This then randomly assign patients in both groups using Microsoft Excel.

- Time study The projected duration of patient recruitment will be adjusted to the rhythm of inclusions to reach 30 patients per group (to follow the normal distribution) or about 6 months of recruitment in the event of observing a strong effect of the tape on the pain.

Acquisition of data:

- Data collected Clinical data for categorization of patients will be identified (age, height (m) Weight (kg), sex).

Investigators will evaluate the postoperative edema by measuring the perimeter of thigh. [6] The perimeter will be measured in millimeters at 1/3 and 2/3 of the distance lateral condyle of the femur - the greater trochanter. The landmarks will be found by palpation and marked for replication, the data measured using a 150 cm graduated Bohin® tape in mm will be performed at the bedside by a student intern in physiotherapy.

To quantify postoperative pain, Investigators use a numerical scale presented in a questionnaire to the patient.

Investigators will note on the last day of patient hospitalization of the amount of analgesic received daily, hang postoperative hospitalization.

- Supports: data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Total hip arthroplasty (THA) anterior approach.

Exclusion Criteria:

* Known allergy to acrylic
* open wounds
* psoriasis,
* skin problems
* On active tumor site,
* lymphedema present before surgery,
* circulatory disorders (phlebitis),
* diabetes with neuropathy,
* not speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of pain on Visual Scale | Day 1
  before then after using the tape

SECONDARY OUTCOMES:
Thigh circumference in centimeters (cm). | Day 1,
  Before then after using the tape

CONTACTS AND LOCATIONS:
Overall Officials: JOUFFROY Pomme, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France